CLINICAL TRIAL: NCT00004423
Title: Controlled Trial of 4-Aminosalicylic Acid in Patients With Small Bowel Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13352; UVTCM-FDR001021
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Crohn Disease; Gastrointestinal Diseases; Rare Diseases | interventions — Aminosalicylic Acid

INTERVENTIONS:
Drug: -aminosalicylic acid

SUMMARY:
OBJECTIVES:

I. Assess the efficacy and safety of 4-aminosalicylic acid in patients with active Crohn's disease of the small bowel.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, placebo controlled, multicenter study. Patients are randomized to receive either oral 4-aminosalicylic acid (4-ASA) or placebo twice a day for 12 weeks. After 12 weeks patients who improved with 4-ASA and those who received placebo are given the option of receiving 4-ASA for an additional year.

Patients who were randomized to receive 4-ASA and continue treatment after 12 weeks are followed every 3 months for 1 year. Patients who were randomized to receive placebo and begin 4-ASA therapy after 12 weeks are followed monthly for 3 months, then every 3 months for 1 year.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Active small bowel Crohn's disease established by clinical evaluation and prior radiologic study, endoscopy, surgical findings and/or histopathology
* Crohn's Disease Activity Index (CDAI) must be between 150 and 450
* No ulcerative or infectious colitis or severe perianal disease

--Prior/Concurrent Therapy--

* Biologic therapy: Not specified
* Chemotherapy: Stable dose of no greater than 20 mg per day of prednisone allowed
* Endocrine therapy: No immunosuppressive drugs within the past 3 months No concurrent immunosuppressive drugs
* Radiotherapy: Not specified
* Surgery: No impending surgery No prior ileostomy or colostomy
* Other: No 5-aminosalicylates within the past 2 weeks No concurrent 5-aminosalicylates No concurrent metronidazol or ciprofloxacin

--Patient Characteristics--

* Age: 18 to 80
* Performance status: Ambulatory
* Hematopoietic: Not specified
* Hepatic: No hepatic disease
* Renal: No renal disease
* Other: Not pregnant (negative pregnancy test required) Fertile patients must use effective contraception No documented salicylate allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1995-12; Study Completion 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: James A. Vecchio, Study Chair — University of Vermont